CLINICAL TRIAL: NCT04885972
Title: A Phase 2, Randomized, Active and Placebo-Controlled, Dose Ranging Study to Evaluate the Efficacy and Safety of Intra-articular Resiniferatoxin to Treat Moderate to Severe Pain From Knee Osteoarthritis
Brief Title: Study to Evaluate Intra-articular Resiniferatoxin to Treat Moderate to Severe Pain From Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTX-OAK-201
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis; Knee Pain Chronic
Keywords: osteoarthritis; knee pain; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — resiniferatoxin; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Resiniferatoxin (Experimental): 7.5 mcg, 10 mcg, 12.5 mcg, 15 mcg, or 20 mcg in 5 mL injected once intra-articularly
  Interventions: Drug: Resiniferatoxin
- Zilretta (Active Comparator): 32 mg in 5 mL injected once intra-articularly
  Interventions: Drug: Zilretta
- Placebo (Placebo Comparator): 5 mL injected once intra-articularly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resiniferatoxin — Resiniferatoxin is a compound purified from natural sources.
  Other Names: RTX
  Arms: Resiniferatoxin
Drug: Zilretta — Zilretta is an extended-release corticosteroid approved to manage osteoarthritis knee pain.
  Other Names: triamcinolone acetonide
  Arms: Zilretta
Drug: Placebo — Vehicle solution
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of a single IA injection of various RTX doses, Zilretta or placebo for the treatment of pain due to moderate to severe osteoarthritis knee pain..

DETAILED DESCRIPTION:
This study is a multi-center, Phase 2, randomized, dose ranging, assessor-blinded, active and placebo-controlled, parallel-group prospective study evaluating the efficacy and safety of a single IA injection of various RTX doses, Zilretta or placebo for the treatment of pain due to moderate to severe osteoarthritis knee pain.

A planned 112 subjects will be randomized to one of 7 groups (n=16 each) with each subject receiving one IA injection in the index knee joint (the knee primarily affected by pain if bilateral).

ELIGIBILITY:
Inclusion Criteria:

* BMI < 50 kg/m
* Have moderate-to-severe pain in the index knee due to osteoarthritis (OA) as assessed by the investigator, based on American College of Rheumatology criteria
* Have had OA pain duration in the index knee ≥ 6 months prior to Screening
* Reports worst daily average pain with walking of ≥ 4 on the 0 to 10 NRS for pain intensity during the week prior to Screening
* Have a knee x-ray or MRI scan with KL grade ≥ 2 in the index knee based upon radiographic images obtained within 3 months prior to Screening (image must be available for review)
* Have had treatment failure with at least two prior analgesic agents (at least one NSAID) defined as discontinuation due to side effects or inadequate response to treatment
* Willing to abstain from other IA injections or knee surgery for at least 6 months after study treatment unless elects early discontinuation from the study
* Able to comply with the study procedures and give informed consent
* If on any analgesic medications, have been taking a stable dose for at least one month prior to screening with no increase in dose leading up to study treatment. Note that if the subject is on "as needed" or PRN analgesic medications, these may be continued during the study
* Willing to follow contraception guidelines

Exclusion Criteria:

* Have a history of a hemorrhagic event that is CTCAEv5 Grade 2 or higher within the 6 months prior to screening
* Have evidence of or history of a serious coagulopathy or hemostasis problem at Screening or Baseline
* Have had an IA injection in the index knee within one month prior to screening (3 months if prior IA injection with Zilretta)
* Have undergone arthroscopic or open surgery or replacement surgery to the index knee within 6 months of screening
* Have surgical hardware or other foreign bodies within the index knee joint
* Have current instability/misalignment in the index knee post repair
* Have a sensory peripheral neuropathy that is CTCAEv5 Grade 2 or higher involving the index leg at Screening
* Have significant pain in other joints or body locations that make it difficult to assess pain in the index knee
* If on opioid analgesics to treat knee OA, have an upper limit of 30 mg/day as converted to an oral morphine equivalent dose
* Have a history of substance abuse
* Have an allergy or hypersensitivity to capsaicin, chili peppers, lidocaine or resiniferatoxin
* Pregnant at Screening or planning on becoming pregnant or currently breastfeeding
* Have had a non-study related minor surgical procedure ≤ 3 days or major surgical procedure ≤ 14 days prior to Screening and must be sufficiently recovered and stable prior to study treatment
* Have any medical condition or medical comorbidities that, in the Investigator's opinion, could adversely impact study participation or safety, conduct of the study, or interfere with pain assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in Worst Average Daily Pain at Week 26 | Baseline to Week 26
  Change from baseline through Week 26 in the weekly mean of Worst Average Daily Pain in the previous 24 hours with walking (WADP) using the Numerical Rating Scale of pain intensity, 0-10 scale (NRS)

SECONDARY OUTCOMES:
Duration of response | Baseline through end of study at Week 52
  Time to return to within 10% of baseline pain score with walking based on the weekly mean WADP scores using the NRS (0-10)
Change in Worst Average Daily Pain at Week 12 | Baseline to Week 12
  Change from baseline through Week 12 in the weekly mean of Worst Average Daily Pain in the previous 24 hours with walking (WADP) using the Numerical Rating Scale of pain intensity, 0-10 scale (NRS).
Change in quality of life | Baseline to Week 26
  Change from baseline to Week 26 in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QoL) subscale
Change in WOMAC score | Baseline to Week 12
  Change from baseline to Week 12 in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score (WOMAC-TW12) and subscale scores

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (6):
- United States (6):
  - Horizon Clinical Research, La Mesa, California
  - Lotus Clinical Research, Pasadena, California
  - Affinity Health, Oak Brook, Illinois
  - Advance Pain, Edgewood, Kentucky
  - HD Research LLC, Bellaire, Texas
  - HD Research LLC, Carrollton, Texas